CLINICAL TRIAL: NCT03668756
Title: Comparison of Computer-Assisted Navigation and Conventional Instrumentation for Bilateral Total Knee Arthroplasty: The Functional Outcome of Mid-Term Follow-up Study
Brief Title: Comparison of Computer-Assisted Navigation and Conventional Instrumentation for Bilateral Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CORPG6G0251
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Arthropathy of Knee Joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Computer-Assisted Navigation TKA: the patients who were received CAS TKA in one limb
  Interventions: Procedure: Computer-Assisted Navigation TKA
- Conventional TKA: the patients who were received conventional TKA in one limb

INTERVENTIONS:
Procedure: Computer-Assisted Navigation TKA — TKAs were performed using the image-free CAS navigation system VectorVision
  Groups: Computer-Assisted Navigation TKA

SUMMARY:
To compare the functional outcomes of Computer-Assisted Navigation (CAS) and Conventional Instrumentation TKA at the 8-year follow-up.

DETAILED DESCRIPTION:
The data of the present study was collected from the review of the medical chart of the patients who were scheduled to undergo staged bilateral TKA and randomly assigned to receive Computer-Assisted Navigation (CAS) TKA in one limb and conventional TKA. Then, comparing the functional outcomes of CAS and Conventional Instrumentation was performed by statistical software.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were scheduled to undergo staged bilateral TKA and randomly assigned to receive CAS TKA in one limb and conventional TKA in the other at the 8-year follow-up.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who were scheduled to undergo staged bilateral TKA and randomly assigned to receive CAS TKA in one limb and conventional TKA in the other at the 8-year follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
International Knee Society (IKS) | up to 8-year follow-up
  To assess the functional outcome of TKA by self-explanatory questionnaire

SECONDARY OUTCOMES:
Radiographic evaluation | Baseline and 3 months after operation
  Standard anteroposterior, lateral radiographs of the knee and standing long-leg radiographs of the lower extremity were obtained pre- and postoperatively. The lower extremities were fully extended so that the tibial tuberosities were facing forward and the lateral malleoli were 15 cm apart to ensure that the tibia was vertical and facing forward with minimal rotation. The X-ray beam (20-25 mA/s; 80-85 kV) was centered at the knee joint level at a distance of 120-140 cm.Radiographic data included the mechanical axis angle and the four component alignments described by Ewald: the femoral valgus (FV) angle; tibial valgus angle (TV); femoral flexion (FF) angle; and tibial flexion angle (TF)
Hospital for Special Surgery (HSS) Questionnaire | Baseline, 8-year follow-up
  To assess the functional outcome of TKA by self-explanatory questionnaire
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Baseline, 8-year follow-up
  To assess the functional outcome of TKA by self-explanatory questionnaire
Short Form-36 (SF-36) Health Survey | Baseline, 8-year follow-up
  To assess the functional outcome of TKA by self-explanatory questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wen-Wei HSU, MD, Principal Investigator — Sports Medicine Center, Chang Gung Memorial Hospital, Chiayi
Locations (1):
- Sports Medicine Center, Chang Gung Memorial Hospital, Pizi, Taiwan

IPD SHARING:
Plan to Share IPD: No